CLINICAL TRIAL: NCT05646459
Title: Effect of Local Cannabidiol on Clinical and Inflammatory Outcomes in Periodontal Maintenance Patients.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was unable to obtain IRB approval because CBD was not legal in Nebraska at that time.
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0217-20-FB
Record Dates: First submitted 2020-04-21; First posted 2022-12-12 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Periodontitis, Adult; Inflammation Gum
MeSH Terms: conditions — Chronic Periodontitis; Gingivitis | interventions — Cannabidiol; Dental Devices, Home Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control - Floss (Placebo Comparator): Subjects will use only floss at study site
  Interventions: Device: floss
- Proxabrush - Control (Sham Comparator): Subjects will use only proxabrush at study site.
  Interventions: Device: proxabrush
- Proxabrush - CBD (Experimental): Subject will use CBD + proxabrush on study site.
  Interventions: Drug: cannabidiol

INTERVENTIONS:
Drug: cannabidiol — This group will locally apply cannabidiol to a posterior, localized 6-9 mm bleeding periodontal pocket.
  Other Names: CBD
  Arms: Proxabrush - CBD
Device: floss — This group will use floss alone at the test site (posterior, localized 6-9 mm bleeding periodontal pocket).
  Arms: Control - Floss
Device: proxabrush — This group will use floss alone at the test site (posterior, localized 6-9 mm bleeding periodontal pocket).
  Other Names: interproximal cleaner
  Arms: Proxabrush - Control

SUMMARY:
This study will determine if cannabidiol (CBD) has any effect on local inflammation in periodontal maintenance patients. Many successful therapies exist for the active, untreated periodontal patient. Unfortunately, periodontology has not yet discovered a therapy that will predictably treat local inflammation in patients who are at risk for further pocketing, bleeding on probing, bone loss and ultimately, tooth loss. Although CBD has been patented in various forms since the 1940s, its acceptance and availability to patients has only recently expanded. Marketing of CBD to periodontal patients as a means to control inflammation is commonplace online and in CBD-specific shops. In determining if CBD is a successful supplement to conventional periodontal inflammation control therapies, millions of patients could benefit from this treatment.

DETAILED DESCRIPTION:
The purpose of this study is to determine if CBD has any effect on local inflammation in periodontal maintenance patients. This research is significant and innovative as it will act as a pivotal study to determine if CBD is worthy of further study in the area of periodontal disease and it will be a human clinical trial focusing on a specific aspect of periodontal disease, the maintenance patient. Many successful therapies exist for the active, untreated periodontal patient. Unfortunately, periodontology has not yet discovered a therapy that will predictably treat local inflammation in these patients which are at risk for further pocketing, bleeding on probing, bone loss and ultimately, tooth loss. Although CBD has been patented in various forms since the 1940s, its acceptance and availability to patients has only recently expanded exponentially. Marketing of CBD to periodontal patients as a means to control inflammation is already commonplace online and in CBD-specific shops; it is the duty of periodontology to determine the efficacy and success of this known anti-inflammatory compound as it relates to clinical periodontal parameters. To determine if CBD is a successful adjunct to conventional periodontal inflammation control therapies would be a boon to the advancement of oral health and to millions of patients that could benefit from this treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic moderate-advanced periodontitis
* one 6-9 mm interproximal probing depth
* overall good systemic health
* history of regular PMT

Exclusion Criteria:

* systemic disease that significantly affect periodontal inflammation and bone turnover
* surgical periodontal therapy in the past year
* pregnant/breast-feeding females.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment Level | baseline
  Amount of epithelial attachment to tooth
Clinical Attachment Level | 6 months
  Amount of epithelial attachment to tooth

SECONDARY OUTCOMES:
Inflammatory Biomarkers | baseline
  IL-1B, IL-10, IL-6
Inflammatory Biomarkers | 6 months
  IL-1b, IL-10, IL-6

CONTACTS AND LOCATIONS:
Overall Officials: Joseph B Bavitz, DMD, Study Chair — UNMC College of Dentistry

IPD SHARING:
Plan to Share IPD: No